CLINICAL TRIAL: NCT06115421
Title: Effect of Low Doses of Hypoxia-inducible Factor- Prolyl Hydroxylase Enzyme Inhibitor Plus Iron in the Treatment of Anemia in Dialysis-dependent Chronic Kidney Disease Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201793
Record Dates: First submitted 2023-10-15; First posted 2023-11-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-04

CONDITIONS: Anemia in Dialysis-dependent CKD Patients
Keywords: Dialysis-dependent CKD patients ,anemia ,hypoxia-inducible factor-; Roxadustatse
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Intervention Model Description: two-arm open-label non randomized active control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral low doses of Roxadustat three times weekly plus iron supplement, (Experimental)
  Interventions: Drug: Roxadustat
- Erythropoiesis-stimulating agents (ESAs) (Active Comparator)
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — hypoxia-inducible factor-prolyl hydroxylase inhibitors (HIF-PHIs)
  Other Names: hypoxia-inducible factor- prolyl hydroxylase enzyme inhibitor

SUMMARY:
this study aims to :

1. To compare the efficacy of combining low doses of Roxadustat Hypoxia-Inducible Factor (HIF)-Prolyl Hydroxylase (PHD) inhibitor and iron versus standard treatment with erythropoietin-stimulating agents (ESA) in the treatment of anemia as a complication of chronic kidney disease (CKD) among dialysis-dependent patients.
2. To emphasize the safety profile of low doses of Roxadustat HIF-PHD.
3. To assess changes in the quality of life of patients with kidney disease before and after treatment.

DETAILED DESCRIPTION:
1- The Ethics Committee of Alexandria University approved conducting the research in April 2023.

2. Informed consent will be obtained from all patients to participate in the trial after a thorough explanation of the nature of the study 3. Dialysis-dependent CKD patients with anemia will be recruited from Alexandria University Hospital &/or private hospitals (if any).

4. Study design: two-arm open-label non randomized active control study 5. Sample size was calculated using G*Power 3, a minimal total hypothesized sample size of 72 eligible adult Dialysis dependent CKD patients (DD -CKD) with anemia [ 36 per group] is needed; taking into consideration 95% confidence level, the effect size of 0.6. and 80% power using a t-test.

6. Three phases will comprise the trial: a screening phase that lasts from 2-4 weeks, a therapy phase that lasts for up to 12 weeks, and a follow-up phase that lasts 2-4 weeks. After obtaining informed consent, during visit 1, we will check the inclusion and exclusion criteria At each visit, the patient's well-being and the occurrence of any Drug-Related Adverse effects (DRAs) will be monitored accurately.

7. The Arabic-translated reliable and valid version of the Kidney Disease Quality of Life questionnaire (KDQOL-36) for patients with CKD will be completed with patients during the interview at the baseline and after fulfilling the whole study period 8. The collected data will be subjected to statistical analysis by the use of suitable techniques to achieve the objectives of the study

ELIGIBILITY:
Inclusion Criteria:

- 1. Ages >18. 2. End Stage Renal Disease (ESRD) on Incident Dialysis (ID), defined as dialysis ≥2 weeks but ≤4 months or stable dialysis (dialysis dependent DD) defined as dialysis for ≥ 4 months &having hemodialysis access.

3. Hb ≤10.5 g/dl during the screening period. 4. Erythropoiesis-stimulating agents (ESAs) naïve patients, ESAs resistant patients, or patients who didn't receive any ESA treatment within 4-6 weeks

Exclusion Criteria:

* 1. Age <18 year or >80 year 2. Known hypersensitivity to active substances, peanuts, soya, or any of the drug excipients.

  3. History of hereditary problems galactose intolerance 4. Systolic BP ≥160 mmHg or diastolic BP ≥95 mmHg, within 2 weeks prior to randomization. Patients may be reevaluated once BP is controlled.

  5. Congestive heart failure (CHF), New York Heart Association (NYHA) Class III or IV 6. Acute coronary syndrome (ACS), a thrombotic/thromboembolic event (eg, deep vein thrombosis (DVT) or pulmonary embolism (PE)), stroke, or seizure, within 12 weeks prior to randomization.

  7. Elective coronary revascularization or elective surgery that is expected to lead to significant blood loss.

  8. Hematologic diseases such as thalassemia, sickle cell anemia, active inflammatory bowel disease, active or chronic gastrointestinal bleeding, significant blood loss, or any other known causes for anemia other than CKD.

  9. Red blood cell transfusion within 6 weeks prior to the first screening visit.

  10. More than one dose of IV iron was received within 12 weeks prior to recruiting.

  11. History of uncontrolled chronic, severe, fulminant, autoimmune, or end-stage liver disease with Aspartate aminotransferase( AST), alanine aminotransferase (ALT) > 3 × upper limit normal (ULN), or total bilirubin > 1.5 × ULN. 12. Any clinically significant inflammatory disorders other than CKD, as any evidence of an active underlying infection, rheumatoid arthritis, systemic lupus, or cancer.

  13. Known and untreated retinal vein occlusion or proliferative diabetic retinopathy, macular degeneration, diabetic macular edema.

  14. Prior organ transplant or a scheduled organ transplantation date. 15. Planning for pregnancy, pregnant, or breastfeeding female patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes in hemoglobin level from baseline | 3 months
  HB g/dl
Iron metabolism parameters change from the baseline | 3 months
  serum iron µg/ml , ferritin µg/l, Total Iron Binding Capacity µg/ml (TIBC) levels, and transferrin saturation (TSAT)%
Safety profile | 3 months
  adverse events will be reported using a pre-prepared checklist

SECONDARY OUTCOMES:
Time to achieve and maintain HB target | 3 months
  desired level (HB) 10-12 g/dL
The need for rescue therapy | 3 months
  1. For the Roxadustat-treated participants (intervention arm) rescue therapy is defined as, red blood cell (RBC) transfusion or erythropoiesis-stimulating agent (ESA).
  2. For erythropoiesis-stimulating agents (ESA) (control arm) rescue therapy is defined as RBC transfusion
The minimum effective dose in combination with iron is needed to achieve the HB target. | 3 months
Change in hepcidin level in the intervention group | 3 months
Change in the Quality of Life (QoL) of the patients after the completion of the study period | 3 months
  Arabic-translated reliable and valid version of the Kidney Disease Quality of Life questionnaire (KDQOL-36) for patients with CKD

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No